CLINICAL TRIAL: NCT05076630
Title: Effect of Air Pollution on Prognosis of Patients With Chronic Obstructive Pulmonary Disease and Its Underlying Biological Mechanism
Brief Title: Air Pollution and Health of COPD Patients
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Furong Deng, Deputy Director of Department of Occupational and Environmental Health Sciences, Peking University
Other Study IDs: IRB00001052-21085
Record Dates: First submitted 2021-09-16; First posted 2021-10-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Air pollution; chronic obstructive pulmonary disease; cardiopulmonary health; biological mechanism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Air Pollutants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Morning urine, exhaled Breath Condensate, saliva and venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Air pollutants — Particulate matter and gaseous pollutants

SUMMARY:
This panel study aims to evaluate the effects of air pollutants on cardiopulmonary health of patients with chronic obstructive pulmonary disease (COPD) and explore the potential biological mechanisms.

DETAILED DESCRIPTION:
This panel study was conducted in a group of stable patients with COPD in Beijing, China. The health measurements including lung function, blood pressure and airway inflammation were conducted, and morning urine, exhaled breath condensate, saliva and venous blood were collected at the time of enrollment and at 3, 6 and 9 months after enrollment. Individual exposures to fine particulate matter (PM2.5), black carbon (BC), ozone (O3) and nitrogen dioxide (NO2) were performed for 24 hours at each follow-up. And the daily concentrations of air pollutants were collected from the Beijing Air Quality Real-time Publishing Platform and meteorological data were collected from the National Meteorological Information Center. The linear mixed effects model was used to analyze the association between air pollution and cardiopulmonary health in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* doctor-diagnosed stable COPD patients
* aged 40 to 80 years
* lived in Beijing for over one year before being recruited
* Agree to participate and sign the informed consent form.

Exclusion Criteria:

* Patients with a history of acute exacerbation in the last 1 month
* Patients with other respiratory diseases such as bronchiectasis and asthma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients aged 40-80 in Beijing, China
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Lung function | Nine months
  Lung function test was conducted.

SECONDARY OUTCOMES:
COPD Assessment Test scores | Nine months
  COPD Assessment Test (CAT) scores were used to assess quality of life in COPD patients on a scale of 0 to 40, with higher scores associated with poorer outcomes.
Modified British Medical Research Council (mMRC) Questionnaire score | Nine months
  Modified British Medical Research Council (mMRC) Questionnaire score was used to assess the severity of dyspnea on a scale of 0 to 4, with a higher score indicating a worse outcome.
ST. George's Respiratory Questionnaire scores | Nine months
  ST. George's Respiratory Questionnaire (SGRQ) scores were used to assess quality of life in patients with COPD on a scale of 0 to 100, with higher scores indicating poorer outcomes.
Blood pressure | Nine months
  Systolic and diastolic blood pressure of participants were measured at least three times by a trained technician.
Respiratory inflammation | Nine months
  Fractional exhaled nitric oxide (FeNO) test was conducted.
Airway and systemic oxidative stress levels | Nine months
  Exhaled Breath Condensate (EBC) and urine samples were collected for oxidative stress analysis.
Systemic inflammation | Nine months
  Venous blood was collected for determination of systemic inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Furong Deng, Doctor, Principal Investigator — Peking University
Locations (1):
- Peking University, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang W, Chen B, Shima M, Zhao C, Guo L, Yoda Y, Li S, Wu S, Chen Y, Guo X, Deng F. PM2.5 as a risk factor for sleep oxygen desaturation in COPD: identifying susceptible individuals by smoking and inflammatory phenotypes. Thorax. 2025 Sep 15;80(10):683-692. doi: 10.1136/thorax-2025-223140. PMID 40541407